CLINICAL TRIAL: NCT00089596
Title: A Safety Study of Infusion of Ex Vivo Selectively Amplified Unrelated Cord Blood Stem Cells in Subjects With Hematological Malignancies Receiving Unrelated Cord Blood Transplantation
Brief Title: Infusion of Specially Treated Umbilical Cord Stem Cells After Chemoradiation Treatment for Blood Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ViaCell (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB001; NCT00301704 (obsolete NCT alias)
Record Dates: First submitted 2004-08-06; First posted 2004-08-10 (Estimated); Last update posted 2007-04-12 (Estimated); Status verified 2007-04

CONDITIONS: Acute Lymphocytic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome; Non-Hodgkin Lymphoma; Chronic Myelogenous Leukemia
Keywords: umbilical cord blood; transplant; ALL; AML; MDS; NHL; CML
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

INTERVENTIONS:
Procedure: Expansion of umbilical cord stem cells

SUMMARY:
This study hopes to show that specially treated umbilical cord cells, called stem cells, can be safely given to a person after they receive chemoradiation therapy or chemotherapy for their illness. During chemoradiation therapy or chemotherapy, a person loses all of the cells that are needed to make the different types of cells in their blood, including their immune system cells. These cells must be replaced in order for the blood and immune systems to work properly. Some people receive bone marrow transplants or other types of stem cell transplants to get the cells they need. CB001 is being developed as an option for people who need bone marrow transplants or other types of transplants to replace those cells. It is also being developed for people who do not have the option of other types of transplants.

ELIGIBILITY:
Inclusion Criteria:

* Do not have identical or 5/6 related matched bone marrow, peripheral blood or umbilical cord
* Stable disease and lack of unrelated donor
* Acute myeloid leukemia (AML) in 2nd or subsequent complete remission or first remission with high risk features
* ALL in 2nd or subsequent remission or first remission with high risk features
* Myelodysplastic syndrome (MDS)
* Non-Hodgkin Lymphoma (NHL)
* Chronic Myelogenous Leukemia (CML)
* Adequate function of heart, liver, kidneys and lungs

Exclusion Criteria:

* Females who are pregnant
* Poor ability to perform daily activities
* Weight under 40 kilograms (88 pounds)
* AML caused by chemoradiation
* Prior stem cell transplant
* Uncontrolled infection at time of transplant
* Active fungal infection
* HIV infection
* Primary myelofibrosis
* Receiving other research drugs
* Unable to provide informed consent

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10
Dates: Start 2004-03; Study Completion 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Gunter, MD, Study Director — ViaCell
Locations (4):
- United States (4):
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York